CLINICAL TRIAL: NCT01653249
Title: A Phase I Clinical Trial of an HPV Therapeutic Vaccine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Arkansas (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 130662; R01CA143130 (NIH)
Record Dates: First submitted 2012-07-26; First posted 2012-07-30 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Human Papillomavirus
Keywords: human papillomavirus (HPV); vaccine; treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- vaccination (Experimental): an escalating dose study of a vaccine consisting of four HPV-16 E6 peptides in combination with Candin® to determine the clinically optimum dose (COD), immunologically optimal dose (IOD), and maximum tolerated dose (MTD). An additional 30 subjects will be vaccinated at the final dose (apparent COD) for further assessment of clinical response.
  Interventions: Biological: Vaccine consisting of four HPV-16 E6 peptides in combination with Candin®

INTERVENTIONS:
Biological: Vaccine consisting of four HPV-16 E6 peptides in combination with Candin®

SUMMARY:
This study will consist of 300 women aged 18-50 years. The study will show that a new therapeutic human papillomavirus (HPV) vaccine designed to regress a precancerous condition called high-grade squamous intraepithelial neoplasia (HSIL)is safe. HPV is known to cause cervical, vaginal, oral, and anal cancers. This novel vaccine will consist of a synthetically made fragment of HPV protein called E6 and yeast extract called Candin®. Previous studies have revealed that immune response to E6 is important in fighting HPV. We also know that injecting Candin has anti-HPV effect since it has been used to treat common warts which are caused by different types of HPV. The current standard treatment for HSIL is loop electrical excision procedure (LEEP). The immune system is the part of the body that fights infection and cancer. This research study will also examine the immune response to the vaccine and its effectiveness in regressing HSIL. Volunteers would be eligible to enroll in the study if they have had a recent Papanicolaou (Pap) smear result indicating HSIL or "Cannot rule out HSIL", and if they meet the inclusion/exclusion criteria. Subjects will be eligible to receive vaccinations if biopsy confirms HSIL. A series of four vaccinations will be given roughly 3 weeks apart, and LEEP will be performed at the end of the study approximately 12 weeks after the last vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-50 years
* Had recent Pap smear result consistent with HSIL or "cannot rule out HSIL" or HSIL on biopsy
* Untreated for HSIL or "Cannot rule out HSIL"
* Able to provide informed consent
* Certain physical exam and blood component parameters within acceptable ranges
* Willingness and able to comply with the requirements of the protocol with a good command of the English language

Exclusion Criteria:

* History of disease or treatment causing immunosuppression (e.g., cancer, HIV, organ transplant, autoimmune disease)
* Being pregnant or attempting to be pregnant within the period of enrollment
* Breast feeding or planning to breast feed within the period of enrollment
* Allergy to Candida antigen
* History of severe asthma requiring emergency room visit or hospitalization
* Current use of beta-blocker medication (may not respond to epinephrine in case of anaphylaxis)
* If in the opinion of the Principal Investigator or other Investigators, it is not in the best interest of the patient to enter this study

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2012-08; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
safety | immediately then up to 7 days post vaccinations
  real-time safety measurement of the combined administration of HPV vaccine and Candin® as measured by dose limiting toxicity as defined by adverse events; safety will be assessed at time of vaccination, 30 minutes post-injection, and daily for 7 days post injections.

SECONDARY OUTCOMES:
clinical and virological/immunological response to the HPV vaccine | within weeks of vaccinations or procedures
  Clinical response as defined by loop electrical excision procedure (LEEP); virological assessment to assess the clearance of HPV infection after vaccination; immunological assessments of T-Cells and circulating immune cells (regulated T-Cells and myeloid derived suppressor cells); and assessment of cervical immune cells.

CONTACTS AND LOCATIONS:
Overall Officials: Mayumi Nakagawa, MD, PhD, Principal Investigator — University of Arkansas; William W Greenfield, MD, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States